CLINICAL TRIAL: NCT04050735
Title: Acute Neural and Immune Effects of Alcohol in People Living With HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1904002429; P20GM130414 (NIH)
Record Dates: First submitted 2019-07-09; First posted 2019-08-08 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2024-10

CONDITIONS: HIV-1-infection; Alcohol Drinking
Keywords: HIV infection; alcohol; brain; inflammation
MeSH Terms: conditions — Alcohol Drinking; HIV Infections; Inflammation | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol, ethyl, moderate dose (Experimental): 0.6 gram ethyl alcohol per kilogram of body weight
  Interventions: Other: Alcohol, ethyl, moderate dose
- Placebo (Placebo Comparator): 0 gram ethyl alcohol per kilogram of body weight
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Alcohol, ethyl, moderate dose — Moderate oral dose of ethyl alcohol
  Arms: Alcohol, ethyl, moderate dose
Other: Placebo — Placebo beverage
  Arms: Placebo

SUMMARY:
This study will examine whether moderate alcohol use in the context of HIV infection exacerbates inflammatory signaling in the immune system and brain. The study will recruit healthy individuals and people living with HIV infection who are otherwise in good health to participate. Participants will complete an experimental protocol that involves controlled alcohol administration and magnetic resonance imaging (MRI). Primary outcomes are plasma biomarkers of inflammation and MRI markers correlated with neuroinflammation. Results will advance understanding of the effects of alcohol use in people living with HIV infection.

DETAILED DESCRIPTION:
A sample of 56 participants, to include equal numbers of people living with HIV and uninfected controls, will be recruited to complete the experimental protocol. Participants will be randomized to one of the two beverage conditions (0.60 g/kg alcohol beverage, 0.00 g/kg placebo beverage). Blood samples will be collected at baseline (prior to beverage administration) and for three hours afterward. Cognitive performance and subjective intoxication will be assessed using standardized measures. MRI scans will be collected 4-5 hours after beverage consumption to capture neurobiological outcomes on the descending limb of blood alcohol.

ELIGIBILITY:
General Inclusion Criteria:

1. 21-60 years old;
2. Able to speak and read English at least at 8th grade level;
3. Alcohol use ≥.60 g/kg at least once in past year. In standard drinks, this amount translates to 1.9-3.0 drinks for an average-weight female and 2.4-3.9 drinks for an average-weight male.
4. Body mass index of 18.5-34.9 kg/m2;
5. Lab tests obtained in past year showing no evidence of acute/chronic Hepatitis B or C infection;
6. HIV-1 serostatus (positive or negative, depending on group) confirmed by standard clinical testing;
7. Able to consume soy and nuts safely (in order to consume the standardized meal).

General Exclusion Criteria:

1. History of heavy drinking on a weekly or more frequent basis, with heavy drinking defined per NIAAA guidelines (≥4 drinks for women, ≥5 drinks for men on a given day), in the past two years;
2. More than five heavy drinking episodes in past 90 days;
3. Seeking or receiving treatment for alcohol/drug use, with exception of smoking cessation treatment;
4. Antibiotic use in past 1 month;
5. Daily use of non-steroidal anti-inflammatory drugs, which are known to increase gut permeability;
6. Disorder of the lower GI tract (e.g., inflammatory bowel disease, ulcerative colitis);
7. Positive urine test for amphetamine, cocaine, methamphetamine, opioids, or benzodiazepines (cannabis use will be assessed but is not an exclusion criterion);
8. Positive screening for past 12-month drug use disorder, indicated by Drug Abuse Screening Test-10 score >2;
9. Current major psychiatric disorder (current major depressive episode, bipolar disorder, psychotic disorder);
10. History of fainting, weakness, infection, excessive bruising, or extreme distress from blood draw;
11. Safety contraindication for MRI (e.g., metal implant); Note: copper intrauterine devices (IUDs) continue to be excluded due to Brown MRI research facility regulations but other non-metal IUDs are allowed;
12. Head trauma with loss of consciousness >10 min;
13. Inability to abstain from nicotine for 8 hours in-session;
14. For cannabis users: inability to abstain for 48 hours prior to study;
15. Pregnant, breastfeeding, or not using effective birth control;
16. Any other clinical condition or therapy that, in the physician's opinion, would make subject unsuitable for study or unable to comply with dosing requirement.

HIV-Specific Inclusion Criteria:

1. On antiretroviral therapy (ART) for ≥6 mos;
2. Labs in past 6 mos showing viral load <100 copies/mL, hemoglobin ≥10.0 g/dL, neutrophil count ≥1,000 cells/μL, and platelet count ≥150,000/μL;
3. No active AIDS diagnosis.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mollie Monnig, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University and The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated by this study will be made available to outside investigators in accordance with NIH guidance and policies on data sharing. Data will be available in summary form and as raw individual-level data for analysis.
Supporting Information: ICF
Time Frame: Individual-level data will be available after papers are accepted for publication.
Access Criteria: Institutions and individuals wishing to access data must contact the Principal Investigator (Peter Monti, PhD). Persons requesting data must do so in writing, identifying the affiliation and how the data will be used. Co-authorship is not required as a condition for receiving data. Users will agree that the recipient must not transfer the data to other users and that the data are only to be used for research purposes. Requestors will be required to sign a data and biospecimen sharing agreement with further stipulations for data use and security.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via online platforms (e.g., social media) and from The Miriam Hospital Infectious Diseases and Immunology Center, the largest outpatient provider of infectious disease treatment in Rhode Island.
Pre-assignment Details: Participants are considered "enrolled" when they provide informed consent for initial screening. However, there is a further eligibility assessment at which participants may be found ineligible for a variety of reasons. Therefore the total number of individuals completing the study is lower than the number of individuals enrolled.
Groups:
- HIV seropositive - placebo group: Individuals with confirmed HIV infection who received the placebo condition
- HIV seronegative - placebo group: Individuals confirmed negative for HIV infection who received the placebo condition
- HIV seropositive - alcohol group: Individuals with confirmed HIV infection who received the alcohol condition
- HIV seronegative - alcohol group: Individuals confirmed negative for HIV infection who received the alcohol condition
Period: Overall Study
Arm/Group | HIV seropositive - placebo group | HIV seronegative - placebo group | HIV seropositive - alcohol group | HIV seronegative - alcohol group
Started | 5 | 15 | 6 | 12
Completed | 5 | 15 | 6 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Seropositive - Placebo Group | HIV Seronegative - Placebo Group | HIV Seropositive - Alcohol Group | HIV Seronegative - Alcohol Group | Total
Number analyzed (Participants) | 5 | 15 | 6 | 12 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (11.1) | 35.73 (11.1) | 40.0 (12.3) | 31.8 (9.4) | 35.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 0 | 5 | 13
  Male | 5 | 7 | 6 | 7 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 5 | 9
  Not Hispanic or Latino | 3 | 15 | 4 | 7 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 3 | 10 | 4 | 7 | 24
  More than one race | 1 | 2 | 1 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 15 | 6 | 12 | 38

OUTCOME MEASURES:

1. Primary Outcome: Plasma Biomarker of Microbial Translocation
Description: Lipopolysaccharide (LPS), measured in pg/ml
Time Frame: 0-3 hours
Population: Data from one participant in the "HIV seronegative - alcohol group" arm was not returned from the analytic laboratory and so this group had 11 rather than 12 participants for the LPS analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | HIV seropositive - placebo group | HIV seronegative - placebo group | HIV seropositive - alcohol group | HIV seronegative - alcohol group
Number analyzed (Participants) | 5 | 15 | 6 | 11
pg/ml
  Hour 0 | 58.562 (26.2243) | 99.285 (48.2314) | 77.232 (31.6189) | 97.343 (42.9950)
  Hour 1 | 52.421 (18.2908) | 91.230 (45.7622) | 81.651 (31.7415) | 98.079 (47.9421)
  Hour 2 | 64.928 (24.6054) | 96.092 (54.8184) | 88.037 (31.6958) | 107.312 (47.1446)
  Hour 3 | 66.267 (25.6505) | 94.090 (50.1699) | 67.979 (14.8000) | 95.877 (50.5859)
Statistical Analysis 1: Comparison: HIV seropositive - placebo group vs HIV seronegative - placebo group vs HIV seropositive - alcohol group vs HIV seronegative - alcohol group; Linear mixed model testing the three-way interaction of HIV serostatus (positive/negative), beverage condition (alcohol/placebo), and time (hour 0, 1, 2, 3); Test type: Other — None of the above apply to this study; p = .343, Mixed Models Analysis; F-test = 1.125

2. Primary Outcome: Plasma Biomarkers of Immune Activation
Description: soluble cluster of differentiation 163 (sCD163), measured in ng/ml
Time Frame: 0-3 hours
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | HIV seropositive - placebo group | HIV seronegative - placebo group | HIV seropositive - alcohol group | HIV seronegative - alcohol group
Number analyzed (Participants) | 5 | 15 | 6 | 12
ng/ml
  Hour 0 | 323.50 (28.333) | 301.22 (94.120) | 376.36 (80.593) | 271.79 (85.204)
  Hour 1 | 261.77 (41.248) | 304.71 (100.360) | 412.88 (95.823) | 276.51 (80.020)
  Hour 2 | 261.51 (45.48) | 298.80 (107.154) | 410.52 (117.886) | 262.46 (87.451)
  Hour 3 | 303.82 (43.385) | 300.68 (105.172) | 405.28 (111.696) | 275.30 (82.670)
Statistical Analysis 1: Comparison: HIV seropositive - placebo group vs HIV seronegative - placebo group vs HIV seropositive - alcohol group vs HIV seronegative - alcohol group; [analysis description as in outcome 1, analysis 1]; Test type: Other — None of the above options apply to this study; p = .026, Mixed Models Analysis; F-test = 3.236

3. Primary Outcome: Cerebral Metabolites
Description: Magnetic resonance spectroscopy will be used quantify cerebral metabolites in brain regions of interest, specifically frontal lobe. Primary metabolites of interest include the summed peak of glutamate and glutamine; choline.
Time Frame: 5 hours
Population: One participant's data was lost due to computational/technical factors.
Measure: Mean (Standard Deviation); unit: mmol/kg of tissue water
Arm/Group | HIV seropositive - placebo group | HIV seronegative - placebo group | HIV seropositive - alcohol group | HIV seronegative - alcohol group
Number analyzed (Participants) | 5 | 14 | 5 | 12
mmol/kg of tissue water
  Glutamate+glutamine | 13.0 (1.5) | 14.6 (5.0) | 12.3 (2.8) | 14.4 (3.2)
  Choline | 1.9 (0.29) | 1.8 (0.38) | 1.75 (0.22) | 1.7 (0.33)
Statistical Analysis 1: Comparison: HIV seropositive - placebo group vs HIV seronegative - placebo group vs HIV seropositive - alcohol group vs HIV seronegative - alcohol group; Test of group by condition interaction on choline; Test type: Other — The above categories do not apply to this type of study; p = .987, ANOVA — The p-value for the interaction of HIV serostatus by beverage condition
Statistical Analysis 2: Comparison: HIV seropositive - placebo group vs HIV seronegative - placebo group vs HIV seropositive - alcohol group vs HIV seronegative - alcohol group; Test of group by condition interaction on summed peak of glutamate plus glutamine; Test type: Other — The above types of tests do not apply to this study; p = .836, ANOVA

4. Primary Outcome: White Matter Diffusivity
Description: Diffusion-weighted MRI will be used to quantify diffusivity metrics in brain white matter. Primary outcome is fractional anisotropy (measured on a scale of 0-1, where 1 reflects total anisotropy).
Time Frame: 5 hours
Population: 2 participants were lost to analysis due to technical/computational reasons.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HIV seropositive - placebo group | HIV seronegative - placebo group | HIV seropositive - alcohol group | HIV seronegative - alcohol group
Number analyzed (Participants) | 5 | 14 | 5 | 12
units on a scale | .560 (.011) | .570 (.009) | .562 (.007) | .574 (.009)
Statistical Analysis 1: Comparison: HIV seropositive - placebo group vs HIV seronegative - placebo group vs HIV seropositive - alcohol group vs HIV seronegative - alcohol group; Test of group by condition interaction on fractional anisotropy (FA); Test type: Other — The above types of tests do not apply to this study; p = .846, ANOVA

5. Secondary Outcome: Subjective Intoxication
Description: Intoxication rating scale (0-10), where a higher rating indicates greater subjective feelings of alcohol intoxication. Participants rate their maximum level of intoxication during the study.
Time Frame: 0-5 hours
Population: Full sample
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIV seropositive - placebo group | HIV seronegative - placebo group | HIV seropositive - alcohol group | HIV seronegative - alcohol group
Number analyzed (Participants) | 5 | 15 | 6 | 12
score on a scale | 1.6 (2.1) | 1.3 (1.5) | 6.0 (1.5) | 5.5 (1.9)
Statistical Analysis 1: Comparison: HIV seropositive - placebo group vs HIV seronegative - placebo group vs HIV seropositive - alcohol group vs HIV seronegative - alcohol group; Test of interaction of group by beverage condition; Test type: Other — The above types of tests do not apply to this study; p = .894, ANOVA

6. Secondary Outcome: Cognitive Functioning
Description: Repeatable Battery for Assessment of Neuropsychological Status standardized scores; Note: this measure was unable to be administered to due coronavirus (COVID-19) pandemic restrictions related to social distancing.
Time Frame: 0-2 hours
Population: Data cannot be reported because this test was not performed. Due to restrictions on human subjects research implemented during the COVID-19 pandemic, researchers were not allowed in the same room as participants for >15 mins total during visits. This test (RBANS) was standardized with the administrator seated at a table across from the test taker. The test takes 20-30 mins to administer. Thus, due to COVID-19 rules, this test could not be administered as standardized.
Arm/Group | HIV seropositive - placebo group | HIV seronegative - placebo group | HIV seropositive - alcohol group | HIV seronegative - alcohol group
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For the duration of a participants' participation (an average of three months from baseline to completion).
Arm/Group | HIV seropositive - placebo group | HIV seronegative - placebo group | HIV seropositive - alcohol group | HIV seronegative - alcohol group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/15 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/15 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 0/5 | 0/15 | 0/6 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT04050735/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT04050735/ICF_001.pdf